CLINICAL TRIAL: NCT05013021
Title: Sprint Interval Training (SIT) on the Endurance, Strength and Velocity Capacities of Healthy Sedentary Subjects
Brief Title: Sprint Interval Training on the Endurance, Strength and Velocity Capacities of Healthy Sedentary Subjects
Acronym: BénéfiSIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20CH238; ANSM (Other: 2021-A01152-39)
Record Dates: First submitted 2021-08-10; First posted 2021-08-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2022-06

CONDITIONS: Sedentary Behavior
Keywords: Sprint Interval Training; VO2max; acute fatigue; chronic fatigue; force-velocity profile
MeSH Terms: conditions — Sedentary Behavior | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Sedentary participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sedentary participants (Other): Series of measures placed throughout the time-course (before, after the 1st , the 2nd and the 3rd block of SIT).
  These measurements consist of physiological measurements (VO2max), neuromuscular capacities (force-speed profile), autonomic nervous system responses (heart rate variability) and blood markers (lactate, CK, cytokinases, µRNA).
  Interventions: Other: Sprint Interval Training

INTERVENTIONS:
Other: Sprint Interval Training — The Sprint Interval Training (SIT) training consists of 3 successive blocks of 5 training sessions each. The sessions are 24 to 48 hours apart.
  . One block lasts two weeks. After the end of one block, the following block begins the day after.
  The Sprint Interval Training lasts 6 weeks.
  Each session consists of a series of sprints, the number of which varies from 8 to 14. Thus a session will last from 30 to 45 min approximately
  So, the time frame of this study is Baseline, Block 1, Block 2 and Block 3 (Not in day or week or month)

SUMMARY:
The present study aims to analyse first, the acute effects generated by a single bout of Sprint Interval Training (SIT) and, secondly, the effects of a long-term intervention on sedentary participants.

DETAILED DESCRIPTION:
The main goal is to determine the optimal dose of high-intensity exercise that enhances the best physiological adaptations.

The cumulative effects of SIT, will be assessed by a series of measures placed throughout the time-course (before, after the 1st , the 2nd and the 3rd block of SIT). Those measures consist of physiological measurements (VO2max), neuromuscular capacities (force-velocity profile) the autonomic nervous system responses (heart rate variability) and blood markers (lactate, Creatine phosphoKinase (CK), cytokinases, µRNA). Acute effects will be measured in the familiarisation sessions (after short (8 sprints) and long (14 sprints) sets) by performing a battery of neuromuscular, perceptual, and autonomic nervous system tests before and after the single session of SIT.

ELIGIBILITY:
Inclusion Criteria:

* untrained healthy (less than 2 hours of sport per week)
* free from muscular, bone or joint injuries
* free from neurologic disease

Exclusion Criteria:

* taking neuroactive substances that can alter corticospinal excitability
* Heart or respiratory failure.
* Subjects who have taken corticosteroids within 3 months (inhalation, infiltration or history of corticosteroid therapy).
* Pregnant woman
* Subject under guardianship

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
oxygen uptake (VO2max) - ml/min/kg | At the end of the 1st, 2nd and 3rd block : Each block = 2 weeks; each block is 1 day apart
  consumption oxygen uptake (VO2max) measured on a cycle ergometer
  The main objective is to determine at which time frame of sprint interval training blocks, the endurance performance (VO2max) is best.

SECONDARY OUTCOMES:
Maximum power (W) | At the end of the 1st, 2nd and 3rd block : Each block = 2 weeks; each block is 1 day apart
  It is measured thanks to the force-speed profile using two sprints of 7s with braking forces of 0 , 4 and 0.7 N.kg-1 respectively.
Maximum theoretical force (N.m) | At the end of the 1st, 2nd and 3rd block : Each block = 2 weeks; each block is 1 day apart
  It is measured thanks to the force-speed profile using two sprints of 7s with braking forces of 0 , 4 and 0.7 N.kg-1 respectively.
Maximum theoretical speed (m/s) | At the end of the 1st, 2nd and 3rd block : Each block = 2 weeks; each block is 1 day apart
  It is measured thanks to the force-speed profile using two sprints of 7s with braking forces of 0 , 4 and 0.7 N.kg-1 respectively.
Maximum isometric force (N.m) | At the end of the 1st, 2nd and 3rd block : Each block = 2 weeks; each block is 1 day apart
  It is measured by means of a voluntary maximum contraction test in which the maximum force generated voluntarily is compared to that voluntarily generated force will be compared to that evoked using electrical stimulation of the femoral nerve.
heart rate variability (HRV) | At the end of the 1st, 2nd and 3rd block : Each block = 2 weeks; each block is 1 day apart
Lactate (mmol/l) | At the end of the 1st, 2nd and 3rd block : Each block = 2 weeks; each block is 1 day apart
  Blood sample
Cytokines (pg/ml) | At the end of the 1st, 2nd and 3rd block : Each block = 2 weeks; each block is 1 day apart
  Blood sample
Creatine Kinase (UI/l) | At the end of the 1st, 2nd and 3rd block : Each block = 2 weeks; each block is 1 day apart
  Blood sample
muscle microRNA | At the end of the 1st, 2nd and 3rd block : Each block = 2 weeks; each block is 1 day apart
  Blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Leonard FEASSON, MD-PhD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lloria-Varella J, Koral J, Ravel A, Murias JM, Feasson L, Busso T. Cardiorespiratory and Neuromuscular Improvements Plateau after 2 wk of Sprint Interval Training in Sedentary Individuals. Med Sci Sports Exerc. 2024 May 1;56(5):876-884. doi: 10.1249/MSS.0000000000003357. Epub 2023 Dec 13. PMID 38109197